CLINICAL TRIAL: NCT06528197
Title: Construction of Clinical Model of Primary Sjogren's Syndrome Combined Traditional Chinese Medicine and Western Medicine Based on Multi-omics
Brief Title: Construction of Clinical Model of Primary Sjogren's Syndrome Combined Traditional Chinese and Western Medicine
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); Beijing Hospital of Traditional Chinese Medicine (Other); Shunyi Hospital, Beijing Traditional Chinese Medicine Hospital (Unknown)
Responsible Party: Principal Investigator, Qingwen Tao, Chief physician, China-Japan Friendship Hospital
Other Study IDs: 2024-1-4065
Record Dates: First submitted 2024-07-12; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Primary Sjögren Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group
- Control group

SUMMARY:
This study aims to establish a large sample cohort of patients with primary sjogren's syndrome, collect multi-omics information of patients with primary sjogren's syndrome, and construct disease diagnosis model and disease prognosis prediction model.

ELIGIBILITY:
Inclusion Criteria:

* Meets the 2002 AECG or 2016 ACR/EULAR classification criteria of primary Sjögren's syndrome.

Exclusion Criteria:

* Comorbid connective tissue disease other than the disease under research.
* Women who are pregnant or breastfeeding.
* Combined severe cardiovascular or cerebrovascular disease, hepatic or renal failure, or severe malignant tumors.
* Other conditions (e.g., cognitive impairment) that the investigators consider ineligible for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary Sjögren's syndrome
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with system involvement | Baseline , 6 months follow-up
  System involvement determined from clinical diagnosis

SECONDARY OUTCOMES:
Mortality | Baseline , 6 months follow-up
  All-cause mortality
Number of participants with tumor | Baseline , 6 months follow-up
  Tumor determined from clinical diagnosis
Number of participants with connective tissue disease | Baseline , 6 months follow-up
  Connective tissue disease determined from clinical diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Jiaqi Chen, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lei C, Zhang X, Zhang Y, Fang Y, Chen J, Liu Z, Zhou X, Tang B, Liao J, Huang Z, Yang J, Wang Z, Liu T, Tao Q, Luo J. Sex differences in primary Sjogren's disease: prognostic impact on mortality and cancer. Biol Sex Differ. 2026 Jan 14. doi: 10.1186/s13293-026-00827-7. Online ahead of print. PMID 41530868